CLINICAL TRIAL: NCT02486705
Title: Pilot Evaluation of PTSD Family Coach, a Mobile Phone App for Family Members of Individuals With PTSD
Brief Title: Evaluation of PTSD Family Coach, a Mobile Phone App for Family Members of Individuals With PTSD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jason Owen, Clinical Psychologist, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 28147
Record Dates: First submitted 2015-04-21; First posted 2015-07-01 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: ptsd; family; caregiver; burden
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PTSD Family Coach Basic (Active Comparator): PTSD Coach basic provides an iOS mobile app with extensive information about caregiving for family members of those with PTSD and additional support resources.
  Interventions: Behavioral: PTSD Family Coach Basic
- PTSD Family Coach Full (Experimental): PTSD Family Coach full provides an iOS mobile app with extensive information about caregiving for family members of those with PTSD, additional support resources, tools for coping with caregiving-related stress, and tools for self-monitoring stress symptoms.
  Interventions: Behavioral: PTSD Family Coach Full

INTERVENTIONS:
Behavioral: PTSD Family Coach Full — PTSD Family Coach mobile app is an iOS mobile phone application designed to provide information, support resources, tools for coping with caregiver-related stress, and tools for self-monitoring stress symptoms.
  Other Names: PTSD Family Coach app- full version
  Arms: PTSD Family Coach Full
Behavioral: PTSD Family Coach Basic — PTSD Family Coach mobile app is an iOS mobile phone application designed to provide information and support resources,
  Other Names: PTSD Family Coach app- basic version
  Arms: PTSD Family Coach Basic

SUMMARY:
The proposed pilot study is designed to test the feasibility, acceptability, and potential effectiveness of a mobile phone application (app) developed by the VA National Center for PTSD (VA NCPTSD) for use by family members of those with Posttraumatic Stress Disorder (PTSD). The primary objective of the proposed study is to assess whether family members of veterans with PTSD find the PTSD Family Coach app to be satisfactory and feasible to use. Secondary objectives are to determine if use of the app increases family members' self-efficacy and their ability to manage their own life stress, which may in part be the result of living with someone who has PTSD.

DETAILED DESCRIPTION:
PTSD Family Coach is a mobile phone app for family members of individuals with PTSD. This application provides:

* education about PTSD
* a self-assessment tool measuring life stress
* self-management skills to address acute distress and stress
* direct connection to support and
* information about VA and community resources for family members of individuals with PTSD

From this research, the investigators wish to learn whether family members of someone with PTSD find the PTSD Family Coach to be satisfactory and feasible to use. The investigators would also like to know if use of the app increases family members' knowledge of PTSD, and its treatment, and their ability to manage their own life stress, which may in part be the result of living with a Veteran with PTSD.

Currently, there are very few resources for family members of Veterans with PTSD. If this research demonstrates that PTSD Family Coach is a promising tool for family members, it has the potential to address a tremendous unmet need using a very cost-effective, scalable solution.

ELIGIBILITY:
Inclusion Criteria:

* currently living with a Veteran with significant PTSD symptoms
* age 18 or older
* own an iPhone, iPad or other iOS compatible device
* currently experiencing at least moderate symptoms of stress

Exclusion Criteria:

* currently enrolled in another study related to PTSD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Caregiver Burden (Montgomery Burden Interview) | 1 month
Stress (Perceived Stress Scale) | 1 month
Use of PTSD Family Coach Mobile App (Study-Specific Survey) | 1 month
Satisfaction with PTSD Family Coach Mobile App (Study-Specific Survey) | 1 month
Depression (PHQ-8) | 1 month
Anxiety (GAD) | 1 month

SECONDARY OUTCOMES:
Stigma Associated with Seeking Mental Health Care (Study-Specific Measure) | 1 month
Perceived Benefits of Mental Health Treatment for PTSD (Study-Specific Measure) | 1 month
Social Constraints (Social Constraints Scale) | 1 month
Partner Self-Efficacy (Study-Specific Measure) | 1 month
Veteran Interest in Treatment for PTSD (Study-Specific Measure) | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto Health Care System, Menlo Park, California, United States

REFERENCES:
- [Derived] van Stolk-Cooke K, Wielgosz J, Hallenbeck HW, Chang A, Rosen C, Owen J, Kuhn E. The PTSD Family Coach App in Veteran Family Members: Pilot Randomized Controlled Trial. JMIR Form Res. 2023 Jan 5;7:e42053. doi: 10.2196/42053. PMID 36602852